CLINICAL TRIAL: NCT04578561
Title: Long-term Follow-up of Prophylactic Mesh Reinforcement After Emergency Laparotomy.
Status: Completed | Type: Observational
Sponsor: José A. Pereira (Other)
Responsible Party: Sponsor-Investigator, José A. Pereira, Jose Antonio Pereira-Rodriguez; M.D; Ph.D., Hospital del Mar
Organization: Hospital del Mar (Other)
Other Study IDs: 20198240I
Record Dates: First submitted 2020-10-05; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Prevention of Incisional Hernia in Emergency Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylactic mesh: Patients who received a prophylactic mesh after emergency surgery due to high risk of incisional hernia.
  Interventions: Procedure: Prophylactic mesh use
- Suture: Patients who's laparotomies closure was using only suture without any abdominal wall reinforcement

INTERVENTIONS:
Procedure: Prophylactic mesh use — After laparotomy sutured clousur the abdominal wall wound is reinforced using a suprafascial synthetic mesh.
  Other Names: Incisional hernia prevention
  Groups: Prophylactic mesh

SUMMARY:
Observational Study analyzing the long-term results of prophylactic mesh used for preventing incisional hernia after emergency midline laparotomies.

DETAILED DESCRIPTION:
Background. Prevention of incisional hernias with a prophylactic mesh in emergency surgery is controversial. The present study aimed to analyze the long-term results of prophylactic mesh used for preventing incisional hernia after emergency midline laparotomies.

Methods. This study was a retrospective analysis of patients who underwent an emergency midline laparotomy between January 2009 and July 2010 with a follow-up period of longer than 2 years. Long-term outcomes and risk factors for the development of incisional hernias between patients who received a prophylactic reinforcement mesh (Group M) and suture (Group S) were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing emergency midline laparotomy

Exclusion Criteria:

* Those with need of concomitant hernia repair.
* Those who received incisions outside the midline.
* Those with delayed abdominal closure.
* Those who died in the immediate postoperative period.
* Those without a minimum 2 years of follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent emergency midline laparotomies in the period between January 2009 and July 2010 in our University Hospital. We included all consecutive patients. with at least 2 years of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Incisional hernia | 2 years
  Detection of clinical or subclinical incisional hernia during postoperative longterm followup

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bravo-Salva A, Argudo-Aguirre N, Gonzalez-Castillo AM, Membrilla-Fernandez E, Sancho-Insenser JJ, Grande-Posa L, Pera-Roman M, Pereira-Rodriguez JA. Long-term follow-up of prophylactic mesh reinforcement after emergency laparotomy. A retrospective controlled study. BMC Surg. 2021 May 18;21(1):243. doi: 10.1186/s12893-021-01243-x. PMID 34006282